CLINICAL TRIAL: NCT00001257
Title: Comparison of Inflammatory Responses in Normal Volunteers and Patients With Abnormal Phagocyte Function Using the Suction Blister Technique
Brief Title: Inflammatory Responses in Normal Volunteers and Patients With Abnormal Immune Responses
Status: Terminated | Type: Observational
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 900120; 90-I-0120
Record Dates: First submitted 1999-11-03; First posted 1999-11-04 (Estimated); Last update posted 2019-08-06 (Actual); Status verified 2019-08-02

CONDITIONS: Healthy Volunteers; Abnormal Phagocyte Function
Keywords: Lymphokines; LTB4; Inflammation; Normal Volunteer; Abnormal Phagocyte Function
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other

SUMMARY:
This study will investigate the inflammatory response. People with abnormal regulation of inflammation and immune defects often have an exaggerated or depressed inflammatory response that results in poor healing of recurrent infections. This study will measure and compare amounts of inflammatory mediators (chemicals involved in the inflammatory response) in healthy normal volunteers and in patients with abnormal immune responses.

Healthy normal volunteers and patients with host defense defects or excessive inflammation, as in vasculitis syndromes, may be eligible for this study. Patients must be between 6 and 65 years of age.

Participants will have eight small blisters raised on the forearm using a gentle suction device. The top of the blisters will be removed with scissors and a plastic template will be placed over the blisters. The wells of the template will be filled with a salt solution or a mixture of the subject s serum (fluid part of the blood without cells) and a salt solution. Some blisters may be covered with coverslips a small round piece of very thin sterilized glass before adding the fluid. Blister fluid will be removed from the wells at 3, 5, 8, and 24 hours with a syringe and analyzed for inflammatory mediators. A scab will form over the blisters and fall off in about 2 weeks.

Participants will have about 4 tablespoons of blood drawn in order to compare the inflammatory mediators in the blood with those in the blister fluid.

DETAILED DESCRIPTION:
Patients with abnormal regulation of inflammation and with host defense defects often have an exaggerated or depressed inflammatory response with resultant difficulty in healing of recurrent infections. Delayed healing can be manifested by either a delay in wound healing, granuloma formation along the incision line, or dehiscence of a partially healed wound without evidence of infection. We are interested in studying the dynamics of host immune defenses during an experimentally induced inflammatory response using a well-studied suction blister device. This protocol is designed to study mediators of inflammation in patients with host defense defects as well as patients with excessive inflammation as in the vasculitis syndromes. We will measure mediators of inflammation (e.g., C5a, leukotriene B4, interleukins, chemokines, tumor necrosis factor, interferon-gamma) by ELISA, radioimmunoassay, High Performance Liquid Chromatography, multiplex cytokine assays, and/or bioactivity assays. Furthermore, molecular characterization and host defense functions (e.g., respiratory burst, chemotaxis, phagocytosis, microbicidal activity) of cells recruited to the blisters will also be examined. In addition to the analysis of cell function, RNA will be prepared and subject to DNA microarray or quantitative RT-PCR studies to measure expression and dynamics of key inflammatory mediators. Many of these factors contribute to the inflammatory process and several are thought to be important in granuloma formation. If patients are found to have abnormal amounts of these mediators when compared to healthy volunteers or patients with other abnormalities it will help us understand the basis for their disease and new therapeutic strategies. For example, this blister study allowed us to identify a patient subsequently shown to have IRAK4 deficiency.

ELIGIBILITY:
* INCLUSION CRITERIA - PATIENTS:

Patients having or thought to have an immune defect between the ages of 6 and 65 years (inclusive) are eligible to participate.

INCLUSION CRITERIA - NORMAL VOLUNTEERS:

Be a healthy adult of either sex and between the ages of 18 and 65 years old.

Weight greater than 110 pounds.

Not have any heart, lung, or kidney disease, or bleeding disorders.

Not have a history of viral hepatitis (B or C) since age 11.

Not have a history of intravenous injection drug use.

Not have a history of engaging in high-risk activities for exposure to the AIDS virus.

Not be pregnant.

EXCLUSION CRITERIA - PATIENTS:

Patients less than 6 or greater than 65 years of age.

EXCLUSION CRITERIA - NORMAL VOLUNTEER:

Less than 18 years old or older than 65 years.

Have viral hepatitis (B or C).

HIV positive.

Receiving chemotherapeutic agent(s), or have underlying malignancy.

Pregnant.

Have history of heart, lung, kidney disease, or bleeding disorders.

Ages: 6 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 169 (Actual)
Dates: Start 1990-04-24; Study Completion 2019-08-02

PRIMARY OUTCOMES:
To identify mediators that contribute to the inflammatory process and granuloma formation by comparing mediators collected from healthy volunteers to patients with abnormal regulation of inflammation and patients with host defense defects. | Ongoing

CONTACTS AND LOCATIONS:
Overall Officials: Kol A Zarember, Ph.D., Principal Investigator — National Institute of Allergy and Infectious Diseases (NIAID)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Dale DC, Wolff SM. Skin window studies of the acute inflammatory responses of neutropenic patients. Blood. 1971 Aug;38(2):138-42. No abstract available. PMID 4933314
- [Background] Hellum KB, Solberg CO. Human leucocyte migration: studies with an improved skin chamber technique. Acta Pathol Microbiol Scand C. 1977 Dec;85C(6):413-23. doi: 10.1111/j.1699-0463.1977.tb03663.x. PMID 343498
- [Background] Kuhns DB, Long Priel DA, Gallin JI. Loss of L-selectin (CD62L) on human neutrophils following exudation in vivo. Cell Immunol. 1995 Sep;164(2):306-10. doi: 10.1006/cimm.1995.1174. PMID 7544694